CLINICAL TRIAL: NCT04118972
Title: In the Mirror: Functional Appreciated Bodies (IM FAB): Piloting an Easily Disseminable Primary Prevention Program
Brief Title: In the Mirror: Functional Appreciated Bodies (IM FAB)
Acronym: IMFAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union College, New York (Other)
Collaborators: University at Albany (Other)
Responsible Party: Principal Investigator, Catherine Walker, Visiting Assistant Professor, Union College, New York
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UnionC
Record Dates: First submitted 2018-10-09; First posted 2019-10-08 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Eating Disorder Symptom; Body Image Disturbance

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two active conditions or a control group.
Who Masked: Investigator
Masking Description: Participants are blinded to their study conditions. Investigators are aware of the study conditions but are not present for or delivering the active portions of the intervention directly. Participants in either active condition receive digitally delivered interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Functionality Mirror Exposure & Journal (Experimental): A text-based functionality gratitude "journaling" prompt three times weekly paired with three weeks of weekly functionality-based guided mirror exposure sessions in the lab (the IM FAB program)
  Interventions: Behavioral: Mirror exposure and text prompt responses
- Pure Mirror Exposure & Gratitude Journal (Active Comparator): Thrice weekly generic (non body-focused) gratitude text prompts and pure mirror exposure in the lab. Participants are not given instructions on how to examine body parts, only instructed to examine the same specific body parts as the Functionality group to control specifically for impacts of the body functionality focus.
  Interventions: Behavioral: Mirror exposure and text prompt responses
- Assessment only control (No Intervention): Assessments at Week 1, Week 3, and 1- and 4-month follow-ups, identical to those received by participants in the active condition

INTERVENTIONS:
Behavioral: Mirror exposure and text prompt responses — Participants in the active interventions have three weekly mirror exposure sessions that are either guided with specific instructions as to where to look and how (only in functionality condition)
  Arms: Functionality Mirror Exposure & Journal; Pure Mirror Exposure & Gratitude Journal

SUMMARY:
The current project aims to examine the concept of promoting attention toward body functionality and gratitude using a weekly functionality-based mirror exposure and body functionality gratitude "journaling" text prompts three days a week for three weeks to examine whether this helps foster positive body image and decrease eating disorder symptoms in a sample of undergraduate females, a population at particularly high risk of body image dissatisfaction and consequent eating disorder development.

DETAILED DESCRIPTION:
Specific Aim 1. First, the project aims to test a gratitude-based body functionality primary prevention program, In the Mirror: Functional Appreciated Bodies (IM FAB), that incorporates mirror exposure with a greater intervention "dose" than that piloted by Brooks and Walker. The increased dose should allow for greater ability for participants to consolidate exposure-based learning. Specifically, more time instructed to appreciate the body's functionality allows for more occasions to redirect critical appearance-oriented cognitions to appreciative, function-based cognitions.

Specific Aim 2. Second, the project aims to pilot test a relatively minimalistic intervention that would be easily translated to app-based delivery format, to help overcome the most-cited barriers to prevention program participation noted by undergraduate students in universal prevention research. Specifically, undergraduate participants who were assigned to a prevention program but did not enroll questioned a need for counseling/therapy, reported preferring to deal with issues on their own, and cited a lack of time as reasons they did not enroll.

Specific Aim 3. Third, the project aims to test this specific functionality mirror exposure approach largely on its own, rather than as part of a multicomponent treatment program, so that its unique contribution in preventing body image dissatisfaction, and ultimately eating disorders, can be assessed. A main goal in prevention and treatment development remains to continuously test components of body-image interventions separately for efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate female aged 18-23 years.

Exclusion Criteria:

* Self-definition as having an active eating disorder
* Participation in the Body Project

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must self-identify as female.
Enrollment: 275 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Multidimensional Body Self-Relations Questionnaire scores (MBSRQ; Cash, 2000) | Change from Baseline MBSRQ scores to 20 weeks
  69-item questionnaire with Likert-type scale ranging from 1-5. Trait body image satisfaction with subscales assessing: Appearance Evaluation, Appearance Orientation, Fitness Evaluation, Fitness Orientation, Health Evaluation, Health Orientation, Illness Orientation, Body Areas Satisfaction, Overweight Preoccupation, and Self-Classified Weight; Scores are averaged for each subscale with a range of 1-5. Fitness, Health, and Appearance Evaluation scores that are higher reflect more positive attitudes about one's fitness, health, and appearance, respectively. Higher appearance, fitness, health, and illness orientation, and overweight preoccupation scores reflect greater investment in appearance, health, concerns about becoming ill, fitness, and preoccupation with weight. Higher Body Areas Satisfaction reflects more positive body image. Higher self-classified weight reflects self-reported higher weight categorization (e.g., overweight or obese)
Change in Eating Disorder Diagnostic Scale scores (EDDS; Stice, Fisher & Martinez, 2004) | Change from baseline EDDS scores to 20 weeks
  Eating disorder diagnostic scale for the DSM-5. This is a diagnostic measure, so participants respond to questions regarding binge eating, purging and other compensatory behaviors, weight and shape concern, weight loss, height, weight, and fear of weight gain to determine whether they meet diagnostic criteria for anorexia nervosa, bulimia nervosa, binge eating disorder, atypical anorexia nervosa, low frequency bulimia nervosa, low frequency binge eating disorder, purging disorder, or night eating syndrome. See http://www.ori.org/files/Static%20Page%20Files/EDDS_5.pdf for specific scoring instructions. Higher scale scores represent greater eating disorder pathology. As a diagnostic tool, respondents need to meet DSM-5 criteria for an eating disorder based on specific item responses, and would be scored as indicating a specific eating disorder diagnosis based on those specific item responses.
Change in Body Checking Questionnaire scores (BCQ; Reas, Whisenhunt, Netemeyer, & Williamson, 2002) | Change from baseline BCQ scores to 20 weeks
  Body checking questionnaire. 23-item 5-point Likert-type scale ranging from 1-5. Three subscales assess: Overall appearance checking, specific body part checking, and idiosyncratic checking. Items are summed for for each subscale and for a total score. Total score ranges from 23-115. Higher scores reflect greater frequency of body checking behaviors.
Change in Body Image Avoidance Questionnaire scores (BIAQ; Rosen, Srebnik, Saltzberg, & Wendt, 1991) | Change from baseline BIAQ scores to 20 weeks
  Body image avoidance questionnaire. Measures avoidance of one's body across a range of evaluative contexts. 19 6-point Likert-type scale ranging from 0-5, with three items reverse scored (12, 13, and 19). Items are summed, with a possible range from 0-95. Higher scores reflect greater body image avoidance and are typically associated with greater psychopathology.
Change in Body Appreciation Scale-2 scores (BAS-2; Tylka, & Wood-Barcalow, 2015) | Change from baseline BAS-2 scores to 20 weeks
  Body appreciation measure. 10-item 5-point Likert-type scale. Items reflect accepting and holding positive views about one's body. Items are averaged with higher scores reflecting great body appreciation.
Change in Functional Appreciation Scale scores (FAS; Alleva, Tylka, & Van Deist, 2017) | Change from baseline FAS scores to 20 weeks
  Scale assesses appreciation of the body's functions. 7-item 5-point Likert-type scale with items ranging from 1-5. Items are averaged with greater scores reflecting greater appreciation of the functions and capabilities of one's body.

SECONDARY OUTCOMES:
Usability Metric for User Experience (UMUX; Finstad, 2010) | Post-Intervention (Week 3)
  4 7-point Likert-type items ranging from 0-6, after recoding, which assesses the usability and ease of the IMFAB protocol. The items are summed for a possible range of 0-24 points, with greater scores representing greater usability of the technology or protocol in question.
Feasibility of mobile application scale, derived from UMUX format | Post-Intervention (Week 3)
  5 7-point Likert-scale items and one open-ended item assessing feasibility of the IMFAB protocol delivery via mobile application. Questions range from 0-6 after recoding and are summed. Greater scores reflect higher ratings of feasibility of adopting IMFAB in mobile application format.
Engagement with IMFAB protocol scale, derived from UMUX format. | Post-Intervention (Week 3)
  9 7-point Likert-type scale items & 3 open-ended questions assessing participant engagement with IM FAB protocol. Likert-type items range from 0-6 and are summed after reverse coding. Greater scores reflect more positive attitudes toward the intervention design (e.g., mirror exposure exercises and gratitude text prompts).

OTHER OUTCOMES:
Gratitude Text Responses - Qualitative | Days 2, 4, 6, 8, 10, and 12
  6 Gratitude text responses during the experimental group intervention period will be assessed with qualitative analyses to assess relationship between responses and primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: D. Catherine Walker, Principal Investigator — Union College
Locations (2):
- United States (2):
  - University at Albany, State University of New York, Albany, New York
  - Union College, Schenectady, New York

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared 6 months after initial publication of data analyses from the current study. Researchers will need to submit a proposal for access to the dataset and demonstrate IRB approval for secondary analysis of the data, if using the dataset for research purposes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after initial publication of data analyses from the current study.
Access Criteria: Researchers will need to submit a proposal for access to the dataset and demonstrate IRB approval if using the dataset for research purposes.

REFERENCES:
- [Background] Cash TF, Fleming EC, Alindogan J, Steadman L, Whitehead A. Beyond body image as a trait: the development and validation of the Body Image States Scale. Eat Disord. 2002 Summer;10(2):103-13. doi: 10.1080/10640260290081678. PMID 16864251
- [Background] Cash TF, Green GK. Body weight and body image among college women: perception, cognition, and affect. J Pers Assess. 1986 Summer;50(2):290-301. doi: 10.1207/s15327752jpa5002_15. PMID 3761129
- [Background] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Background] Reas DL, Whisenhunt BL, Netemeyer R, Williamson DA. Development of the body checking questionnaire: a self-report measure of body checking behaviors. Int J Eat Disord. 2002 Apr;31(3):324-33. doi: 10.1002/eat.10012. PMID 11920995
- [Background] Alleva JM, Tylka TL, Kroon Van Diest AM. The Functionality Appreciation Scale (FAS): Development and psychometric evaluation in U.S. community women and men. Body Image. 2017 Dec;23:28-44. doi: 10.1016/j.bodyim.2017.07.008. Epub 2017 Aug 17. PMID 28822275
- [Background] Stice E, Telch CF, Rizvi SL. Development and validation of the Eating Disorder Diagnostic Scale: a brief self-report measure of anorexia, bulimia, and binge-eating disorder. Psychol Assess. 2000 Jun;12(2):123-31. doi: 10.1037//1040-3590.12.2.123. PMID 10887758
- [Background] Stice E, Fisher M, Martinez E. Eating disorder diagnostic scale: additional evidence of reliability and validity. Psychol Assess. 2004 Mar;16(1):60-71. doi: 10.1037/1040-3590.16.1.60. PMID 15023093
- [Background] Froh JJ, Fan J, Emmons RA, Bono G, Huebner ES, Watkins P. Measuring gratitude in youth: assessing the psychometric properties of adult gratitude scales in children and adolescents. Psychol Assess. 2011 Jun;23(2):311-24. doi: 10.1037/a0021590. PMID 21443367

DOCUMENTS (1):
  • Informed Consent Form (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT04118972/ICF_000.pdf